CLINICAL TRIAL: NCT06223646
Title: A Phase 1/2a Study to Evaluate the Safety, Tolerability, Preliminary Efficacy, and Pharmacokinetic Characterization of KQ-2003 for Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: A Study of KQ-2003 CAR-T Cell Therapy for Patients With Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novatim Immune Therapeutics (Zhejiang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KQ-2003-AC101
Record Dates: First submitted 2023-12-22; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase 1: Low dose group (Experimental): Infusion of KQ-2003 CAR T-cells by single dose of 1.0×10^6 CAR-T cells/kg
  Interventions: Biological: KQ-2003 CAR T-cells
- Phase 1: Medium dose group (Experimental): Infusion of KQ-2003 CAR T-cells by single dose of 2.0×10^6 CAR-T cells/kg
  Interventions: Biological: KQ-2003 CAR T-cells
- Phase 1: High dose group (Experimental): Infusion of KQ-2003 CAR T-cells by single dose of 3.0×10^6 CAR-T cells/kg
  Interventions: Biological: KQ-2003 CAR T-cells
- Phase 2a: RP2D (Experimental): After all subjects in the Phase 1 dose-escalation study completed DLT observation, RP2D was determined based on the analysis results for the phase 2a expansion study.
  Interventions: Biological: KQ-2003 CAR T-cells

INTERVENTIONS:
Biological: KQ-2003 CAR T-cells — KQ-2003 CAR T-cell therapy involves autologous chimeric antigen receptor T-cells, capable of targeting both human B cell maturation antigen (anti-BCMA CAR) and CD19 antigen molecules (anti-CD19 CAR) simultaneously as a cellular therapy.

SUMMARY:
This is a multicenter, open-label, dose-escalation/expansion phase 1/2a study to evaluate the safety, tolerability, pharmacokinetic/pharmacodynamic characteristics and determine the recommended dose of KQ-2003 CAR T-cells for patients with Relapsed/Refractory Multiple Myeloma

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, male or female;
* Diagnosis of MM with relapsed or refractory disease;
* Eastern Cooperative Oncology Group (ECOG) Performance ≤2 ;
* Expected survival of at least 12 weeks;
* Participant has measurable disease;
* Adequate venous access for the apheresis of peripheral blood mononuclear cell;
* Adequate organ function;
* Able and willing to comply with the study protocol and follow-up plan, and sign the informed consent form in writing.

Exclusion Criteria:

* Received any treatment that might influence the activity of CAR-T cells prior to the collection of peripheral blood mononuclear cells;
* Have history of vaccination within the 4 weeks preceding the collection of peripheral blood mononuclear cells;
* Have active bleeding or venous thromboembolic events requiring anticoagulation;
* Have tested positive for cytomegalovirus and/or mycobacterium tuberculosis, or had any uncontrolled active infection within 14 days prior to the collection of peripheral blood mononuclear cells;
* Subjects infected with active HBV or HCV, HIV, syphilis;
* Subjects with known central nervous system disease or multiple myeloma involving the central nervous system (CNS) or presenting with CNS-related symptoms;
* Patients currently experiencing active autoimmune diseases;
* Diagnosed with immunodeficiency or receiving any other form of immunosuppressive therapy within 7 days prior to enrollment in this study.
* Have following severe diseases: unstable angina, cerebrovascular accident or transient ischemic attack, myocardial infarction , New York Heart Association (NYHA) Class ≥ III, congestive heart failure, poorly controlled severe arrhythmias or other cardiac diseases requiring mechanical support; subjects with known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal; subjects with known moderate or severe persistent asthma, or a history of asthma within the past 2 years, or currently having any category of uncontrolled asthma; subjects requiring oxygen to maintain adequate oxygen saturation; subjects with hypertension whose blood pressure cannot be lowered to the following range despite treatment with two or more antihypertensive medications;.
* Subjects with malignancies other than multiple myeloma;
* Have any non-hematologic toxicity resulting from prior treatments that cannot be restored to ≤ grade 1 or baseline, excluding alopecia and grade 2 neuropathy;
* History of alcohol abuse, drug addiction, substance abuse, or mental illness within the past year;
* Presence of acute graft-versus-host disease (GVHD) or extensive chronic GVHD of Grade ≥ 2 requiring treatment within the 4 weeks before enrollment, or as judged by the investigator to likely require anti-GVHD treatment during the study; Subjects who had previously received BCMA-CD19 dual-target CAR-T cell products or autologous stem cell transplantation within 12 weeks before the collection of peripheral blood mononuclear cells;
* Known allergy or hypersensitivity reactions to cyclophosphamide, fludarabine, dimethyl sulfoxide (DMSO), CD19, or BCMA-targeted drugs;
* Subjects had participated in other clinical trials and used its investigational drugs within the 3 months prior to the collection of peripheral blood mononuclear cells
* Pregnant or lactating women
* Any situation that the investigator believes may increase the risk of subjects or interfere with the results of clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose-limiting toxicity (DLT) | Within 28 days of receiving KQ-2003 CAR T-cells transfusion therapy
  For DLT evaluation, severity (grade) is classified according to common terminology criteria for adverse events version 5.0 (CTCAE v5.0).
Maximum Tolerated Dose (MTD) | Within 28 days of receiving KQ-2003 CAR T-cells transfusion therapy
  At least 6 subjects in the MTD dose group must complete the DLT assessment.
Adverse Event | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Safety will be assessed by adverse events (AEs), which include clinically significant abnormalities identified during a medical test (e.g. laboratory tests, electrocardiogram, vital signs, physical examinations). AEs will be coded by Medical Dictionary for Regulatory Activities (MedDRA) and their severity will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE, version 5.0).
Recommended Phase 2 Dose (RP2D) | Through study completion, an average of 1 year
  To determine after all subjects in the Phase 1 dose-escalation study completed DLT observation
Objective response rate (ORR) | Through study completion, an average of 2 years
  The definition of ORR is the proportion of subjects achieving sCR, CR, VGPR, or PR confirmed by efficacy reassessment after a minimum interval of three months. ORR is calculated as (sCR+CR+VGPR+PR) divided by the total number of cases, multiplied by 100%.

SECONDARY OUTCOMES:
Stringent complete response rate (sCRR) | Through study completion, an average of 2 years
  The definition of sCRR is the proportion of subjects achieving sCR confirmed by efficacy re-assessment after a minimum interval of three months.
Duration of Response (DOR) | Through study completion, an average of 2 years
  DOR will be calculated among responders from the date of initial documentation of a response to the date of first documented evidence of progressive disease.
Disease Control Rate (DCR) | Through study completion, an average of 2 years
  The proportion of subjects achieving sCR, CR, VGPR, PR, MR, or disease stability (SD) confirmed by efficacy reassessment after a minimum interval of three months is defined as the DCR.
Progression-free Survival (PFS) | Through study completion, an average of 2 years
  The time interval from the first administration of the investigational drug to the first observation of disease progression is calculated, considering the date of entry for patients who died for reasons other than disease progression before progression occurred.
Overall Survival (OS) | Through study completion, an average of 2 years
  OS is the time from the start of cell infusion to the death of the subject.
Microscopic Residual Disease (MRD) Negativity Rate and Duration | Through study completion, an average of 2 years
  The duration of MRD negativity is the period during which both bone marrow MRD and imaging remain negative.
Maximum concentration (Cmax) | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Blood and bone marrow samples will be collected and used for pharmacokinetics assessments.
Time to maximum plasma concentration (Tmax) | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Blood and bone marrow samples will be collected and used for pharmacokinetics
Levels of IL-6 | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Blood samples will be collected and used for pharmacodynamic to evaluate the levels about cytokine levels
Levels of IFN-γ | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Blood samples will be collected and used for pharmacodynamic to evaluate the levels about cytokine levels
CD4+T lymphocyte count | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Blood samples will be collected and used for pharmacodynamic to evaluate the levels about peripheral blood lymphocyte subsets
CD8+T lymphocyte count | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  Blood samples will be collected and used for pharmacodynamic to evaluate the levels about peripheral blood lymphocyte subsets
ADA | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  The trial will evaluate the positive rate, titer and duration or persistence of ADA following the administration of CAR T-Cells.
Nab | Minimum 2 years after KQ-2003 CAR T-cells infusion (Day 1)
  The trial will evaluate the positive rate, titer and duration or persistence of Nab following the administration of CAR T-Cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College Hospital, Beijing, China